CLINICAL TRIAL: NCT01369706
Title: Safety of Screening Procedures With Hand-held Metal Detectors Among Patients With Implanted Cardiac Rhythm Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GER-EP-007
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Electromagnetic Interference
Keywords: electromagnetic interference; hand-held metal detector; pacemaker; cardioverter-defibrillator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hand-held metal detector (Other): Exposure to two hand-held metal detectors
  Interventions: Device: Hand-held metal detector

INTERVENTIONS:
Device: Hand-held metal detector — 2 different hand-held metal detectors: (1) PD 140 (CEIA S.p.A., Arezzo, Italy) and (2) MH 5 (Vallon GmbH, Eningen, Germany)

SUMMARY:
Patients with implanted pacemaker (PM) or cardioverter-defibrillator (ICD) systems are restrained in daily life by possible electromagnetic interference (EMI). Case reports suggest EMI between PM or ICD systems and hand-held metal detectors that are intensively used as part of security screening processes in e.g. airport controls.

The objective was to determine the safety of screening procedures for ferrous materials with regard to possible in vivo EMI between hand-held metal detectors and PM and ICD systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for routine pacemaker or cardioverter defibrillator control
* appropriate PM/ICD function

Exclusion Criteria:

* atrial or ventricular sensing abnormalities that could not be avoided by reprogramming of device parameters
* low battery status of the device such as elective replacement indicator (ERI)
* intrinsic heart rate > 120 beats per minute (bpm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Jilek, MD, Principal Investigator — Deutsches Herzzentrum München; Christof Kolb, MD, Study Chair — Deutsches Herzzentrum München
Locations (2):
- Deutsches Herzzentrum München, München, Germany
- Cardiology Department, Hospital "Henry Dunant", Athens, Greece

REFERENCES:
- [Result] Jilek C, Tzeis S, Vrazic H, Semmler V, Andrikopoulos G, Reents T, Fichtner S, Ammar S, Rassias I, Theodorakis G, Weber S, Hessling G, Deisenhofer I, Kolb C. Safety of screening procedures with hand-held metal detectors among patients with implanted cardiac rhythm devices: a cross-sectional analysis. Ann Intern Med. 2011 Nov 1;155(9):587-92. doi: 10.7326/0003-4819-155-9-201111010-00005. PMID 22041947

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hand-held Metal Detector
Started | 388
Completed | 388
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hand-held Metal Detector
Number analyzed (Participants) | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 295
Region of Enrollment [Number; unit: participants]
  Greece | 71
  Germany | 317

OUTCOME MEASURES:

1. Primary Outcome: Electromagnetic Interference
Description: inhibition of the pacemaker, loss of capture, inappropriate mode switch, ventricular oversensing, power-on-reset, device reprogramming or loss of function
Time Frame: time during exposure to hand-held metal detector (2x 30 sec)
Population: Electromagnetic interference
Measure: Number; unit: participants
Arm/Group | Hand-held Metal Detector
Number analyzed (Participants) | 388
participants | 0

ADVERSE EVENTS:
Arm/Group | Hand-held Metal Detector
Serious Adverse Events (participants affected / at risk) | 0/388
Other Adverse Events (participants affected / at risk) | 0/388

LIMITATIONS AND CAVEATS:
Convenience sample of patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes